CLINICAL TRIAL: NCT05958277
Title: Vitamin B12 vs B3 for Nerve Regeneration and Functional Recovery After Pediatric Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KRL Hospital, Islamabad (Other)
Responsible Party: Principal Investigator, Hassan Mumtaz, Principal Researcher, KRL Hospital, Islamabad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRL/02/19/2
Record Dates: First submitted 2023-06-30; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Niacinamide; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B3 (Experimental): Vitamin B3 group
  Interventions: Drug: Vitamin B3
- Vitamin B12 group (Experimental): Vitamin B12 group
  Interventions: Drug: Vitamin B12

INTERVENTIONS:
Drug: Vitamin B3 — Vitamin B3 upto 16 mg/day
  Arms: Vitamin B3
Drug: Vitamin B12 — Vit B12 upto 250 mcg per day
  Arms: Vitamin B12 group

SUMMARY:
A traumatic brain injury (TBI) is among the most frequent reasons for neurological impairment in young people. The investigators investigated whether vitamin B12 vs B3 therapy could reduce the severity of traumatic brain injury (TBI) due to their positive effects on axon regrowth following nerve damage. The method utilized was a series of non-random samples. With a 95% confidence interval and a 5% margin of error, a total sample of 300 patients was estimated using Epi Info. Participants in our study comprised both boys and girls with severe TBI ages 6 to 15 years old.

Two groups of 300 children were recruited. B3 (16 mg/day) was administered to group 1 and B12 (125-250 mcg/day) was provided to group 2. It is evaluated through follow-ups on a range of tests to evaluate cognitive capacity, sensorimotor activity and staircase test (working and reference memory). Pre-and post-treatment GCS measurements were conducted. Three weeks and a year following the treatment of TBI, children underwent neurobehavioral testing. The measurement of gait analysis was done. The standard error and mean of statistically examined data were shown by paired t-test.

DETAILED DESCRIPTION:
A traumatic brain injury (TBI) is among the most frequent reasons for neurological impairment in young people. The investigators investigated whether vitamin B12 vs B3 therapy could reduce the severity of traumatic brain injury (TBI) due to their positive effects on axon regrowth following nerve damage. The method utilized was a series of non-random samples. With a 95% confidence interval and a 5% margin of error, a total sample of 300 patients was estimated using Epi Info. Participants in our study comprised both boys and girls with severe TBI ages 6 to 15 years old.

Two groups of 300 children were recruited. B3 (16 mg/day) was administered to group 1 and B12 (125-250 mcg/day) was provided to group 2. It is evaluated through follow-ups on a range of tests to evaluate cognitive capacity, sensorimotor activity and staircase test (working and reference memory). Pre-and post-treatment GCS measurements were conducted. Three weeks and a year following the treatment of TBI, children underwent neurobehavioral testing. The measurement of gait analysis was done. The standard error and mean of statistically examined data were shown by paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 15 years old
* Children with severe TBI of
* Children of both genders

Exclusion Criteria:

* Those with mild injury
* Stable Glasgow Coma Scale
* Not willing to consent

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Stair Climb Test (SCT) score | 18 months
  The stair test is a measurement of functional strength, balance, and agility achieved by ascending and descending a specific number of steps. Scoring involves recording the total time taken to ascend and descend the steps to the nearest 100th of a second. Lower values indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- KRL Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided